CLINICAL TRIAL: NCT03854175
Title: Effect of Vaginal Sildenafil Citrate on Endometrial Preparation and Outcome in Frozen Thawed Embryo Transfer Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 51
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sildenafil Citrate; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil group (Active Comparator): 40 women are give sildenafil citrate 25mg vaginally every 6 hours (a half of 50 mg tablet is crushed and dissolved in 2cc of distilled water and injected in to vagina) starting from day 2-14 of the cycle, in addition to oral 2mg of estradiol valerat 6-8 hourly from the day 2-14 of the menstrual cycle
  Interventions: Drug: sildenafil citrate; Drug: Estradiol Valerate 2 MG
- estradiol group (Active Comparator): 40 women are given oral estradiol valerate tablets 2mg 6-8 hourly from the day 2-14 of the cycle to prepare the endometrium in addition to placebo in the same way as sildenafil
  Interventions: Drug: Estradiol Valerate 2 MG

INTERVENTIONS:
Drug: sildenafil citrate — 25mg vaginally every 6 hours (a half of 50 mg tablet is crushed and dissolved in 2cc of distilled water and injected in to vagina) starting from day 2-14 of the cycle
  Arms: Sildenafil group
Drug: Estradiol Valerate 2 MG — 2mg 6-8 hourly from the day 2-14 of the cycle to prepare the endometrium

SUMMARY:
A total of 80 Patients who meet these conditions will enter the study and be divided into two groups based on randomized tables.

To prepare the endometrium,

Group A : 40 women are given oral estradiol valerate tablets 2mg 6-8 hourly from the day 2-14 of the cycle to prepare the endometrium

Group B : 40 women are give sildenafil citrate 25mg vaginally every 6 hours (a half of 50 mg tablet is crushed and dissolved in 2cc of distilled water and injected in to vagina) starting from day 2-14 of the cycle, in addition to oral 2mg of estradiol valerat 6-8 hourly from the day 2-14 of the menstrual cycle . Estrogen and progesterone (prontogest 400mg pessaries ) are given 3 days prior to embryo transfer. Sildenafil is discontinued 48-72 hours prior to the embryo transfe due sildenafil may have some detrimental effects on endometrium in the implantation window

DETAILED DESCRIPTION:
A total of 80 Patients who meet these conditions will enter the study and be divided into two groups based on randomized tables.

To prepare the endometrium,

Group A : 40 women are given oral estradiol valerate tablets 2mg 6-8 hourly from the day 2-14 of the cycle to prepare the endometrium

Group B : 40 women are give sildenafil citrate 25mg vaginally every 6 hours (a half of 50 mg tablet is crushed and dissolved in 2cc of distilled water and injected in to vagina) starting from day 2-14 of the cycle, in addition to oral 2mg of estradiol valerat 6-8 hourly from the day 2-14 of the menstrual cycle . Estrogen and progesterone (prontogest 400mg pessaries ) are given 3 days prior to embryo transfer. Sildenafil is discontinued 48-72 hours prior to the embryo transfe due sildenafil may have some detrimental effects on endometrium in the implantation window.

For assessing endometrial vascularity (on day 14 of cycle), two dimension power Doppler characteristics as normal quality of color, color gain-3.4, pulse repetition frequency of 600Hz and wall motion filter of 50Hz are applied in all examinations. By following Applebaum's zones of vascularity for categorizing endometrial vasculaity: Zone 1 vascularity-When blood vessls reach the hypoechoic endometrio-myometria junction, Zone 2 vascularity when the vessels reach the outer hyperechoic line of en-dometrium, Zone 3 vascularity when it reach the intervening hypoechoic area, Zone 4 vascularity when the vessels are seen reaching the central echogenic line .

After 5 days when the endometrial pattern is triple line pattern (trilaminar) and endometrial thickness is more than 8mm,embryos will be transferred. All patients have a luteal phase support by giving a daily doses of estradiol valerat 2mg oral daily and 100mg progesterone (prontogest 100mg ampoule ) as an intramuscular which will be continued two weeks after the em-bryos transfer. In case BHCG is tested and proved to be positive, estradiol valerat and progesterone are continueed until the 11th week of pregnancy. Then, four weeks after the embryo transfer, the number of gestational sacs are determined by vaginal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing their first frozen embryo transfer cycle.
* have at least two high quality frozen embryos

Exclusion Criteria:

* 1. a history of endocrine diseases. 2. a history of hysteroscopic surgeries. 3. cardiovascular, renal and liver diseases. 4. hypotension (blood pressure <90/50 mmHg). 5. a history of stroke or myocardial infarction.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness | At the day of embryo transfer
  ultrasound measurement of the endometrial thickness at the fundus

SECONDARY OUTCOMES:
Endometrial vascularity | At the day of embryo transfer
  two dimension power Doppler characteristics as normal quality of color, color gain-3.4, pulse repetition frequency of 600Hz and wall motion filter of 50Hz are applied in all examinations. By following Applebaum's zones of vascularity for categorizing endometrial vasculaity: Zone 1 vascularity-When blood vessls reach the hypoechoic endometrio-myometria junction, Zone 2 vascularity when the vessels reach the outer hyperechoic line of en-dometrium, Zone 3 vascularity when it reach the intervening hypoechoic area, Zone 4 vascularity when the vessels are seen reaching the central echogenic line
clinical pregnancy rate | 4 weeks after embryo transfer
  detection of intrauterine gestational sac by transvaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided